CLINICAL TRIAL: NCT04767789
Title: Double-blind, Placebo-controlled, Randomized Pilot Clinical Trial to Evaluate the Efficacy and Safety of the Probiotic Strains Limosilactocillus Reuteri DSM 32910 and Lacticaseibacillus Paracasei DSM 32851 on Glucose Homeostatis in Prediabetic Adults
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of the Probiotic Strains Limosilactocillus Reuteri DSM 32910 and Lacticaseibacillus Paracasei DSM 32851 on Glucose Homeostatis in Prediabetic Adults
Acronym: NOVOGLUCOSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Novozymes A/S (Industry)
Collaborators: Biofortis, Merieux NutriSciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PEC20022; 2021-A00210-41 (Other: ID-RCB Number); 295204 (Other: IRAS Project ID)
Record Dates: First submitted 2021-02-04; First posted 2021-02-23 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Prediabetic State; Dysglycemia
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NZ-GHMH-01 (Experimental): Dietary supplement in shape of capsule to be taken once per day in the evening.
  Interventions: Dietary Supplement: NZ-GHMH-01
- Placebo (Placebo Comparator): The placebo is in shape of capsule to be taken once per day in the evening and in which only the active ingredients are not present.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: NZ-GHMH-01 — Each randomized subject will consume 1 capsule daily bringing 100 mg (≥ 2 x 109 CFU) of active ingredient during 16 weeks (from V2 to V5 visits).
  Arms: NZ-GHMH-01
Dietary Supplement: Placebo — Each randomized subject will consume 1 capsule with no active ingredient daily during 16 weeks (from V2 to V5 visits).
  Arms: Placebo

SUMMARY:
The aim of this international, randomized, parallel arms, double-blind, placebo-controlled clinical trial is to investigate the safety and efficacy of a combination of the two Lactobacillus strains (NZ-GHMH-01) on glucose and insulin metabolism, in prediabetic subjects. This trial will include prediabetic (insulin resistant) subjects with excessive body weight (over-weight or obese, showing abdominal or visceral obesity) to be able to investigate the effect of the probiotic NZ-GHMH-01 on glycaemic control.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 75 years (limits included)
* Having BMI between 18,5 and 40 kg/m² (limits included)
* Prediabetic
* For women: Non menopausal with the same reliable contraception or menopausal without or with hormone replacement therapy
* Agreeing to keep his lifestyle habits unchanged throughout the study
* With stable weight within ± 5% in the last three months
* Having a good general and mental health with in the opinion of the investigator
* Having signed informed consent form
* Affiliated with a social security scheme (for French sites only)
* Agreed to be registered on the subjects in the "VRB" (biomedical research file (for French sites only))
* Having HbA1c level ≥ 5.7% and ≤ 6.4%

Exclusion Criteria:

* Metabolic disorder such as diabetes or uncontrolled thyroidal trouble or other metabolic disorder;
* Having a history of medication for diabetes and dyslipidemia
* Uncontrolled hypertension
* Severe chronic disease or gastrointestinal disorders
* Having done the second injection of COVID-19 vaccination or between the first and the second injection within the last 2 weeks prior to V1 visit
* Food allergy or intolerance or hypersensitivity to any of the study products' ingredient
* Pregnant or lactating women or intending to become pregnant within 3 months ahead
* Smoking subject (more than 5 cigarettes per day)
* Having a history of bariatric surgery
* Having a history of any surgery in the 3 months before V1 visit or having scheduled any surgery within 6 months ahead
* Under dietary supplement except fibers, omega 3 and vitamins (other than Vitamin D3) if the subject agrees to keep his/her intake unchanged throughout the study;
* Under treatment which could significantly affect parameter(s) followed during the study
* Under antibiotic treatment in the 3 to 6 months before V1 visit
* With significant change in food habits or in physical activity in the 3 months before V1 visit or not agreeing to keep them unchanged throughout the study
* With a current or planned in the next 5 months specific diet (hyper or hypocaloric, vegan…) or putted in place since less than 3 months before the inclusion visit
* With a personal history of anorexia nervosa, bulimia or significant eating disorders according to the investigator
* Abuse of alcohol, defined as more than 21 alcohol units per week for men and 14 units for women, or unwillingness to refrain from alcohol intake the day before V2 and V5 visits
* Having a lifestyle deemed incompatible with the study according to the investigator
* Taking part in another clinical trial or having taken part in another clinical trial in the 3 months before the inclusion visit;
* Having received, during the last 12 months, indemnities for clinical trial higher or equal to 4500 Euros (for French sites only);
* Under legal protection (guardianship, wardship) or deprived from his rights following administrative or judicial decision;
* Presenting a psychological or linguistic incapability to sign the informed consent;
* Impossible to contact in case of emergency.
* Having blood ASAT, ALAT or GGT levels out of range and clinically significant according to the investigator
* Having CBC with hemoglobin < 11 g/L or leucocytes < 3000 /mm3 or leucocytes > 16000 /mm3 or clinically significant abnormality according to the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2022-11-29 (Actual); Study Completion 2022-11-29 (Actual)

PRIMARY OUTCOMES:
Glycated Hemoglobin A1c (HbA1c) | V2 (randomization) and V5 (16 weeks of intervention)
  Change from Baseline of HbA1c level between V2 and V5 visits (in %) between both groups.

SECONDARY OUTCOMES:
Glycated Hemoglobin A1c (HbA1c) | V3 (4 weeks of intervention), V4 (12 weeks of intervention) and V5 (16 weeks of intervention)
  Change from baseline of HbA1c level
Glucose kinetic parameters: ΔPeak and Cmax | V2 (randomization) and V5 (16 weeks of intervention)
  Change from baseline of ΔPeak (g/L) and Cmax (g/L)
Glucose kinetic parameters: T max | V2 (randomization) and V5 (16 weeks of intervention)
  Change from baseline of T max (min)
Incremental Area Under the Curve (iAUC) of glucose | V2 (randomization) and V5 (16 weeks of intervention)
  Change from baseline of the value of the iAUC of glucose, obtained during OGTT (iAUC0-120min)
Incremental Area Under the Curve (iAUC) of insulinemia | V2 (randomization) and V5 (16 weeks of intervention)
  Change from baseline of the value of the iAUC of insulinemia, obtained during OGTT (iAUC0-120min)
Homeostasis Model of Assessment - insulin resistance (HOMA-IR) | V2 (randomization), V3 (4 weeks of intervention), V4 (12 weeks of intervention) and V5 (16 weeks of intervention)
  Change from baseline of HOMA-IR index
Quantitative Insulin sensitivity Check Index (QUICKI) | V2 (randomization), V3 (4 weeks of intervention), V4 (12 weeks of intervention) and V5 (16 weeks of intervention)
  Change from baseline of QUICKI index
Insulin Sensitivity Index (ISI) | V2 (randomization), V3 (4 weeks of intervention), V4 (12 weeks of intervention) and V5 (16 weeks of intervention)
  Change from baseline of ISI index
Fasting Plasma Glucose (FPG) | V2 (randomization), V3 (4 weeks of intervention), V4 (12 weeks of intervention) and V5 (16 weeks of intervention)
  Change from baseline of FPG levels
Fasting insulinemia | V2 (randomization), V3 (4 weeks of intervention), V4 (12 weeks of intervention) and V5 (16 weeks of intervention)
  Change from baseline of fasting insulinemia levels
Glycemia | V2 (randomization) and V5 (16 weeks of intervention)
  Change from baseline of glycemia level
Glucagon Like Peptide 1 (GLP-1) | V2 (randomization) and V5 (16 weeks of intervention)
  Change from baseline of GLP-1 level
Weight | V2 (randomization), V3 (4 weeks of intervention), V4 (12 weeks of intervention) and V5 (16 weeks of intervention)
  Change from baseline of weight(in kg)
Body Mass Index (BMI) | V2 (randomization), V3 (4 weeks of intervention), V4 (12 weeks of intervention) and V5 (16 weeks of intervention)
  Change from baseline of BMI (in kg/m2)
Waist and Hip | V2 (randomization), V3 (4 weeks of intervention), V4 (12 weeks of intervention) and V5 (16 weeks of intervention)
  Change from baseline of Waist measurement (in cm) and Hip Circumference (in cm)
Anthropometric ratios | V2 (randomization), V3 (4 weeks of intervention), V4 (12 weeks of intervention) and V5 (16 weeks of intervention)
  Change from baseline of Waist to Hip ratio and Waist to Height ratio
Liver function | V2 (randomization), V3 (4 weeks of intervention), V4 (12 weeks of intervention) and V5 (16 weeks of intervention)
  Change from baseline of Aspartate Amino Transferase (ASAT), Alanine Amino Transferase (ALAT) and Gamma Glutamyl Transpeptidase (GGT) levels (expressed in ukat/L)
Total bilirubin | V1 (screening) and V5 (16 weeks of intervention)
  Change from baseline of Total bilirubin levels (expressed in umol/L)
Triglycerides | V2 (randomization), V3 (4 weeks of intervention), V4 (12 weeks of intervention) and V5 (16 weeks of intervention)
  fasting blood concentrations of triglycerides (expressed in g/L)
Lipid homeostasis | V2 (randomization), V3 (4 weeks of intervention), V4 (12 weeks of intervention) and V5 (16 weeks of intervention)
  fasting blood concentrations of total cholesterol, High Density Lipoprotein cholesterol (HDLc), non-HDLc and Low Density Lipoprotein cholesterol (LDLc) (expressed in mmol/L)
high-sensitivity C-reactive Protein (CRPhs) | V2 (randomization), V3 (4 weeks of intervention), V4 (12 weeks of intervention) and V5 (16 weeks of intervention)
  Change from baseline of the CRPhs
Cytokines | V2 (randomization), V3 (4 weeks of intervention), V4 (12 weeks of intervention) and V5 (16 weeks of intervention)
  Change from baseline of the Cytokines IL-1alpha, IL-1beta, IL-6, IL-10, IL-12p70 and monocyte chemoattractant protein 1 (MCP1)
Tumor Necrosis Factors alpha (TNFα) | V2 (randomization), V3 (4 weeks of intervention), V4 (12 weeks of intervention) and V5 (16 weeks of intervention)
  Change from baseline of the TNFα
Overall health | V2 (randomization), V3 (4 weeks of intervention), V4 (12 weeks of intervention) and V5 (16 weeks of intervention)
  Change from baseline of participant overall health (evaluated with SF36 questionnaire)
Blood metabolites | V2 (randomization) and V5 (16 weeks of intervention)
  Change from baseline of Cholic acid, Chenodeoxycholic acid, Deoxycholic acid, Lithocholic acid, Ursodeoxy cholic acid, Taurocholic acid and Glycochenodeoxycholic acids
Gastrointestinal Symptoms | V2 (randomization), V3 (4 weeks of intervention), V4 (12 weeks of intervention) and V5 (16 weeks of intervention)
  Change from baseline of gastrointestinal symptoms (evaluated with Gastrointestinal Symptom Rating Scale)

OTHER OUTCOMES:
Incidence of adverses events | V1 (Inclusion), V2 (randomization), V3 (4 weeks of intervention), V4 (12 weeks of intervention) and V5 (16 weeks of intervention)
  Incidence of adverses events
Heart Rate | V1 (Inclusion), V2 (randomization), V3 (4 weeks of intervention), V4 (12 weeks of intervention) and V5 (16 weeks of intervention)
  overall health through hemodynamic parameters: Heart Rate (expressed in bpm)
Blood pressure | V1 (Inclusion), V2 (randomization), V3 (4 weeks of intervention), V4 (12 weeks of intervention) and V5 (16 weeks of intervention)
  overall health through hemodynamic parameters: Systolic Blood Pressure and Diastolic Blood Pressure (expressed in mmHg)
Complete Blood Count (CBC) | V1 (Inclusion), V2 (randomization), V3 (4 weeks of intervention), V4 (12 weeks of intervention) and V5 (16 weeks of intervention)
  overall health through CBC: Leukocytes, Red blood cells, Hemoglobin, Hematocrit, Poly. Neutrophils, Poly. Neutrophils, Poly. Eosinophils, Poly. Eosinophils, Poly. Basophils, Poly. Basophils, Lymphocytes, Lymphocytes, Monocytes, Monocytes, Platelets (expressed in Giga/L and %)
Fecal zonulin | V2 (randomization) and V5 (16 weeks of intervention)
  Change from baseline of fecal zonulin level
Fecal calprotectin | V2 (randomization) and V5 (16 weeks of intervention)
  Change from baseline of fecal calprotectin level

CONTACTS AND LOCATIONS:
Locations (8):
- France (2):
  - Clinical Investigation Unit Biofortis, Saint-Herblain, Pays de la Loire Region
  - Clinical Investigation Unit Paris, Paris
- Romania (5):
  - Neomed Brasov, Brasov
  - Fundatia Ana Aslan International, Bucharest
  - Military Hospital- Spitalul Militar Central Dr "Carol Davila", Bucharest
  - Parhon Institute- Institutul National de Endocrinologie C.I. Parhon, Bucharest
  - Suceava County Hospital - Spitalul Județean de Urgență "Sfântul Ioan cel Nou", Suceava
- CPS Research, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No